CLINICAL TRIAL: NCT06791629
Title: Pulsed Field Ablation Versus Radiofrequency Ablation for Persistent Atrial Fibrillation: A Randomized, Open-label, Non-inferior Study
Brief Title: Pulsed Field Ablation Versus Radiofrequency Ablation for Persistent Atrial Fibrillation
Acronym: PRAISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-PeAF ablation
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Persistent Atrial Fibrillation; Radiofrequency Catheter Ablation; Pulsed Field Ablation
Keywords: persistent atrial fibrillation; Radiofrequency Catheter Ablation; pulsed field ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency Ablation (Active Comparator)
  Interventions: Device: Radiofrequency Ablation
- Pulsed Field Ablation (Experimental)
  Interventions: Device: Pulsed Field Ablation

INTERVENTIONS:
Device: Pulsed Field Ablation — Patients will be treated with pulsed field ablation for atrial fibrillation.
  Arms: Pulsed Field Ablation
Device: Radiofrequency Ablation — Patients will be treated with radiofrequency ablation for atrial fibrillation.
  Arms: Radiofrequency Ablation

SUMMARY:
This clinical trial aims to compare the efficacy and safety of pulsed field ablation and radiofrequency ablation to treat persistent atrial fibrillation in adults.

Participants will:

Undergo pulsed field ablation or radiofrequency ablation. Keep follow-up for at least 12 months.

DETAILED DESCRIPTION:
Traditional treatment options for persistent atrial fibrillation (PeAF) include pharmacological management, electrical cardioversion, and catheter ablation. Pulmonary vein isolation (PVI) has become the cornerstone of ablation therapy and has been shown to be effective in clinical practice. However, its efficacy is relatively limited in patients with persistent AF compared with those with paroxysmal AF, and many patients still experience recurrence after treatment.

In recent years, linear ablation strategies based on alcohol ablation have been shown to improve the one-year maintenance of sinus rhythm in patients with PeAF. Traditional radiofrequency ablation (RF) has demonstrated good outcomes but still has certain limitations when dealing with PeAF. In several clinical studies, pulsed field ablation (PFA), an emerging and innovative technique, has shown non-inferiority in treating paroxysmal AF. Furthermore, PFA has also demonstrated significant efficacy in linear ablation sites such as the mitral isthmus line, posterior left atrial wall, and tricuspid isthmus line, highlighting its potential in treating PeAF. This study aims to compare the safety and efficacy of PFA and radiofrequency ablation (RF) in the treatment of PeAF through a multi-center, prospective, randomized, open-label, non-inferiority clinical trial, to provide a safer and more effective treatment option for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years
* Patients with non-valvular persistent atrial fibrillation undergoing their first catheter ablation (AF duration: 3 months to 3 years)
* Left atrial diameter on parasternal long-axis view of echocardiogram < 50 mm
* Agree to be randomly assigned to the ablation strategy and able to follow up

Exclusion Criteria:

* Atrial fibrillation due to reversible causes
* LVEF < 30%
* Severe congenital heart disease
* Severe liver or kidney dysfunction (eGFR < 15, Child-Pugh grade 3), or history of dialysis
* History of cardiac surgery, such as coronary artery bypass grafting, mechanical valve or prosthetic valve replacement
* History of pacemaker implantation, left atrial appendage closure, or patent foramen ovale closure
* Contraindications to oral anticoagulation
* Contraindications to right or left heart catheterization
* Pregnancy
* Life expectancy < 1 year (e.g., advanced malignancy, end-stage renal disease)
* Currently enrolled in another trial evaluating medical devices or drugs
* Other situations where the investigator determines the subject is unsuitable for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Freedom from any documented atrial arrhythmia lasting for >30s in the absence of antiarrhythmic therapy in 12 months after the index ablation procedure (excluding a blanking period of 3 months) | From the end of the 3-month blanking period post-ablation to the 12-month follow-up

SECONDARY OUTCOMES:
Freedom from any documented atrial arrhythmia in 12 months after the index ablation procedure | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Freedom from any documented atrial fibrillation lasting for >30s in 12 months after the index ablation procedure (excluding a blanking period of 3 months) | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Freedom from any documented atrial tachycardia and atrial flutter episodes in 12 months after the index ablation procedure | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Freedom from any documented atrial arrhythmia in the absence of antiarrhythmic therapy in 12 months after multiple ablation procedure (excluding a blanking period of 3 months) | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
The atrial fibrillation burden (percentage of time) monitored over 12 months | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Cardiovascular-related hospitalizations in 12 months after the index ablation procedure | From the end of the 3-month blanking period post-ablation to the 12-month follow-up
Perioperative complications in 30 days after the index ablation procedure | From the end of the ablation to the 30 days follow-up
  Cardiac tamponade or perforation, permanent phrenic nerve palsy, acute coronary artery occlusion, stroke/thromboembolism/transient ischemic attack, pulmonary vein stenosis, left atrial-esophageal fistula, vascular complications requiring intervention (e.g., pseudoaneurysm, arteriovenous fistula), coronary artery spasm, renal failure due to hemolysis, death, and other treatment-related complications requiring intervention or prolonging hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No